CLINICAL TRIAL: NCT06011811
Title: Cluster Headache Treatment Survey
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Clusterbusters, Inc. (Unknown)
Responsible Party: Principal Investigator, Mark J Burish, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-23-0212
Record Dates: First submitted 2023-08-19; First posted 2023-08-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with episodic or chronic cluster headache: Patients with a diagnosis of episodic or chronic cluster headache, as diagnosed by a health care professional and to be confirmed by questions on the study survey.

SUMMARY:
The objective of this study is to survey patients with cluster headache about treatment effectiveness and their views on treatments. Participants will complete one brief questionnaire online.

ELIGIBILITY:
Inclusion Criteria:

* Patients with episodic or chronic cluster headache that has been diagnosed by a health care professional (no documentation is needed, participant must simply state that he or she has been diagnosed)

Exclusion Criteria:

* Unable to speak English (the survey is only in English)
* Unable to use a computer to take the online survey
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is patients with episodic or chronic cluster headache that has been diagnosed by a health care professional. The cluster headache diagnosis will be verified via the survey using a validated cluster headache diagnostic screen.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of cluster headache treatment as assessed by a survey | at the time of survey completion, expected to be 6-12 months

SECONDARY OUTCOMES:
Opinions on new cluster headache treatment as assessed by a survey | at the time of survey completion, expected to be 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Burish, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study survey — https://survey.alchemer.com/s3/7134634/Cluster-Headache-Medication-Psychedelic-Use-Survey-2023